CLINICAL TRIAL: NCT05273866
Title: A Technological Intervention in Pain Control on Intravenous Cannulatıon in Children Virtual Reality Glasses: A Randomized Controlled Study
Brief Title: The Effect of Virtual Reality Glasses on Pain on Intravenous Cannulatıon in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Haci Bektas Veli University (Other)
Responsible Party: Principal Investigator, Bahriye Kaplan, Principal Investigator, Nevsehir Haci Bektas Veli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 84902927
Record Dates: First submitted 2022-02-08; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Pain, Procedural
Keywords: distraction; intravenous cannulation; pain; school-aged children; virtual reality glasses
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Virtual reality video application
  Interventions: Other: Virtual reality
- control group (No Intervention): control group

INTERVENTIONS:
Other: Virtual reality — Virtual Reality video application reduces pain by distracting. The intervention group was watched video during the procedure, starting before the procedure.
  Arms: Virtual reality

SUMMARY:
This study was carried out to determine the effect of virtual reality glasses on reducing pain during vascular access in children. The study consisted of 70 children (35 children in the virtual reality video group and 35 children in the control group). Ethics committee approval, permissions from institutions and informed voluntary consent of the children were obtained in order to conduct the study. The data of the study were collected with Child Descriptive Characteristics Form, Parent Descriptive Characteristics Form, Visual Analog Scale (VAS), Revised Facial Expression Pain Scale (FPS-R), Intervention Monitoring Form, Child Behavior Observation Form and Parent Behavior Observation Form. In the study, the children in the experimental group were shown a video with virtual reality glasses during the vascular access procedure. Before and after the study; The child and his parents were asked to evaluate the pain experienced/will experience during the procedure, the children's heart rate, O2 saturation, body temperature were measured, and the behaviors of the child and the parent during the procedure were evaluated. A p value of <0.05 was considered statistically significant in data analysis.

DETAILED DESCRIPTION:
This randomized controlled experimental study was conducted to determine the effect of virtual reality glasses on reducing pain during vascular access in children. The study was conducted among children aged 7-12 years in a tertiary hospital. Children in the experimental group (n=35) and control group (n=35); Age, gender, class of education, previous hospitalization and vascular access experience criteria were selected similar (p>0.05). Data were collected with Child Descriptive Characteristics Form, Parent Descriptive Characteristics Form, Visual Analog Scale (VAS), Revised Facial Expression Pain Scale (FPS-R), Intervention Monitoring Form, Child Behavior Observation Form, and Parent Behavior Observation Form. In the study, the children in the experimental group were shown a video with virtual reality glasses during the vascular access procedure. Before and after the study; The child and his parents were asked to evaluate the pain experienced/will experience during the procedure, the children's heart rate, O2 saturation, body temperature were measured, and the behaviors of the child and the parent during the procedure were evaluated. Data were used post-power analysis, descriptive statistics, Shapiro Wilk, Pearson chi-square, Mann Whitney U and Two-Related-Samples Tests. A p value of <0.05 was considered statistically significant in data analysis.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 7-12,
* Does not have a disease that causes chronic pain,
* Not taking any analgesic medication in the last 8 hours before the procedure,
* No mental or neurological disability,
* Having no visual or auditory problems that prevent you from applying the scales or watching videos,
* Does not have eye problems and/or does not use glasses to be able to wear VR glasses,
* The first vascular access procedure was performed during this hospitalization at the clinic,
* Vascular access opened on the first try,
* Speaking and understanding Turkish,
* Children whose parents and themselves agreed to participate in the study were included in the study.

Exclusion Criteria:

* Does not understand the Turkish language
* the child is under 7 years old or 12 years older
* having vision, hearing or speech problems
* having a mental or neurological disability

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS), Change: | 2 minutes before and 2 minutes after Intravenous Cannulatıon
  The severity of the pain marked by the child on the scale ranges from 0 to 10. If the severity increases after the procedure, it indicates that the pain increases, and if it decreases, it indicates that the pain decreases.
Faces Pain Scale-Revised (FPS-R), Change: | 3 minutes before and 3 minutes after Intravenous Cannulatıon
  In the scale consisting of facial expressions, each facial expression has a number equivalent. The severity of pain marked by the child on the scale ranges from 0 to 10. If the severity increases after the procedure, it indicates that the pain increases, and if it decreases, it indicates that the pain decreases.

SECONDARY OUTCOMES:
Physiological parameters | 2 minutes before and 2 minutes after Intravenous Cannulatıon
  Heart Rate, Change
Physiological parameters | 3 minutes before and 3 minutes after Intravenous Cannulatıon
  Oxygen saturation, Change

CONTACTS AND LOCATIONS:
Overall Officials: Bahriye Kaplan, Doctor, Study Director — Nevsehir Haci Bektas Veli University
Locations (1):
- Bahriye Kaplan, Nevşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No